CLINICAL TRIAL: NCT05558969
Title: The Effect of Prophylactic Magnesium Use in Pregnant Women on Reversal of Neuromuscular Block With Sugammadex:Evaluation With TOF
Brief Title: The Effect of Magnesium Use in Reversal of Neuromuscular Block With Sugammadex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Meryem Onay, assistant professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESOGU 4
Record Dates: First submitted 2022-09-01; First posted 2022-09-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2022-09

CONDITIONS: Magnesium Sulfate; Pregnancy; Pre-Eclampsia; Neuromuscular Blockade
Keywords: Preeclampsi; Magnesium sulfate; Sugammadex
MeSH Terms: conditions — Toxemia | interventions — Sugammadex

STUDY DESIGN:
Intervention Model Description: A total of 30 pregnant women, who are taking magnesium and not taking magnesium, will be included in the study to be taken by cesarean section under general anesthesia.At the end of surgery, whether sugammadex reverses the effect of NMBA will be evaluated. The time up to TOF 0.9 will be recorded.A blood sample will be taken to measure simultaneous calcium and magnesium values.
Who Masked: Participant, Investigator
Masking Description: It will be evaluated by another investigator (blind) who does not know in which group the patient is using magnesium sulfate during the intraoperative period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregnant women taking magnesium (Active Comparator): The patient group who received magnesium as a 4-6 g loading and 2-3 g/h maintenance dose to prevent convulsions in preeclampsia. Pregnant will be operated under general anesthesia
  Interventions: Drug: pregnant women taking magnesium
- control group (Placebo Comparator): Pregnant will be operated under general anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregnant women taking magnesium — The patient group who received magnesium as a 4-6 g loading and 2-3 g/h maintenance dose to prevent convulsions in preeclampsia. Pregnant will be operated under general anesthesia. Sugammadex 4mg/kg will be administered when TOF 0 response is seen at the end of surgery. The time from TOF 0 to TOF 0.9 will be recorded. Magnesium and calcium levels in the blood will be studied.
  Other Names: magnesium level and sugammadex
  Arms: pregnant women taking magnesium
Drug: Placebo — Pregnant women who do not receive magnesium therapy and who will be operated under general anesthesia. Sugammadex 4mg/kg will be administered when TOF 0 response is seen at the end of surgery. The time from TOF 0 to TOF 0.9 will be recorded. Magnesium and calcium levels in the blood will be studied.
  Other Names: magnesium level and sugammadex
  Arms: control group

SUMMARY:
Magnesium therapy used for seizure prophylaxis in patients with preeclampsia. Magnesium has been shown to prolong the effect of nondepolarizing neuromuscular blocking agents (NMBA) and neostigmine used to reverse the effect of NMBA in general anesthesia . In this study, the investigators aimed to evaluate time from sugammadex injection to Train-of-four ratio 0.9 who receieved magnesium therapy in reversing the effect of neuromuscular blocking agent during the recovery period and the relationship between magnesium level and duration of action of sugammadex

DETAILED DESCRIPTION:
Rapid-onset and short-acting agents should be preferred in induction, and full induction doses should be applied since they do not receive premedication and increased volume of distribution. Rapid serial induction and intubation should be performed in pregnancies greater than 20 weeks due to the risk of aspiration. Magnesium potentiates and prolongs the effect of nondepolarizing neuromuscular blocking agents. It is recommended that the TOF value be between 0 and 2 for adequate muscle relaxation in cesarean section anesthesia. In anesthesia induction; thiopental 3-6mg/kg, rocuronium 1mg/kg, and fentanyl 1mcg/kg and dormicum 2mg will administered after the baby birth. Sevoflurane 2-3% and 50% oxygen + 50% air are used for maintenance. If TOF is 0, sugammadex 4mg/kg will be administered to reverse the effect of the muscle relaxant.A blood sample will be taken to measure simultaneous calcium and magnesium values. Patients with a TOF ≥0.9 (gold standard for extubation) or patients will be clinically evaluated and the decision to extubate will be made.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are scheduled for cesarean section under general anesthesia (pregnant women who do not use magnesium) and who use magnesium for prophylaxis in preeclampsia.

Exclusion Criteria:

* Eclampsia,
* chronic hypertension,
* connective tissue disorder,
* muscle disease, neurological problems,
* thyroid dysfunction,
* kidney disease, heart disease,
* patients with severe allergic reaction to the agents to be used,
* sepsis,
* hypovolemia, abruptio placenta, placenta previa,
* conditions that will prolong the effect of muscle relaxants (drug use ),
* pregnant women who did not want to be included in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant
Enrollment: 30 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Recovery time | at end of surgery (Postoperative 2 hours)
  TOF 0.9 Achieving Time and evaluate the relationship between blood magnesium and calcium level with sugammadex effect.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Onay, asst. prof., Principal Investigator — Eskisehir Osmangazi University Faculty Of Medicine
Locations (1):
- Eskisehir Osmangazi Universıty Faculty of Medicine, Eskişehir, Eski̇şehi̇r, Turkey (Türkiye)

REFERENCES:
- [Background] Czarnetzki C, Tassonyi E, Lysakowski C, Elia N, Tramer MR. Efficacy of sugammadex for the reversal of moderate and deep rocuronium-induced neuromuscular block in patients pretreated with intravenous magnesium: a randomized controlled trial. Anesthesiology. 2014 Jul;121(1):59-67. doi: 10.1097/ALN.0000000000000204. PMID 24608361
- [Background] Chattopadhyay S, Das A, Pahari S. Fetomaternal outcome in severe preeclamptic women undergoing emergency cesarean section under either general or spinal anesthesia. J Pregnancy. 2014;2014:325098. doi: 10.1155/2014/325098. Epub 2014 Apr 17. PMID 24864211
- [Background] Stourac P, Adamus M, Seidlova D, Pavlik T, Janku P, Krikava I, Mrozek Z, Prochazka M, Klucka J, Stoudek R, Bartikova I, Kosinova M, Harazim H, Robotkova H, Hejduk K, Hodicka Z, Kirchnerova M, Francakova J, Obare Pyszkova L, Hlozkova J, Sevcik P. Low-Dose or High-Dose Rocuronium Reversed with Neostigmine or Sugammadex for Cesarean Delivery Anesthesia: A Randomized Controlled Noninferiority Trial of Time to Tracheal Intubation and Extubation. Anesth Analg. 2016 May;122(5):1536-45. doi: 10.1213/ANE.0000000000001197. PMID 26974018